CLINICAL TRIAL: NCT02262481
Title: A Randomized, Double Blinded, Placebo Controlled Trial of Oral Progestogen Supplementation in the Prevention of Recurrent Uterine Contraction in Preterm Labor
Brief Title: Oral Progestogen Supplementation in the Prevention of Recurrent Uterine Contraction in Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Vorapong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RA57/104
Record Dates: First submitted 2014-10-03; First posted 2014-10-13 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dydrogesterone (Active Comparator): tocolytic + corticosteroids + Dydrogesterone 10 mg/tablet prepare in capsule, 1 cap oral every 12 hours, starting form enrollment until gestational age 37 weeks
  Interventions: Drug: dydrogesterone
- Placebo (Placebo Comparator): tocolytic + corticosteroids + Placebo prepare in capsule, 1 cap oral every 12 hours, starting form enrollment until gestational age 37 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dydrogesterone
  Other Names: Duphaston
  Arms: Dydrogesterone
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of oral progesterone supplementation in preterm labor on the prevention of recurrent uterine contraction and prolonging pregnancy period, and its side effect.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Preterm labor
* GA24-34wk
* Intact membranes

Exclusion Criteria:

* Maternal/fetal condition requiring immediate delivery ex. Chorioamnionitis, fetal distress
* Placenta previa
* medical and obstetric complications
* allergy to dydrogesterone

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The recurrence of uterine contraction within 48 hours after stop tocolytic | 48 hours

SECONDARY OUTCOMES:
Time from preterm labor pain to delivery | 9 weeks
Gestational age at delivery | 9 weeks
Number of newborn with respiratory distress syndrome | 9 weeks
side effects | 9 weeks
Number of newborn with intraventricular hemorrhage | 9 weeks
Number of newborn with necrotizing enterocolitis | 9 weeks
Number of newborn with sepsis | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Preterm birth. In: Cunningham FG, Leveno KJ, Bloom SL, Hault JC, Rouse DJ, Spong CY, editors. Williams Obstetrics. 23rd ed. McGraw-Hill; 2010. p. 804-831.
- [Background] American College of Obstetricians and Gynecologists; Committee on Practice Bulletins-Obstetrics. ACOG practice bulletin no. 127: Management of preterm labor. Obstet Gynecol. 2012 Jun;119(6):1308-17. doi: 10.1097/AOG.0b013e31825af2f0. PMID 22617615
- [Background] Committee on Practice Bulletins-Obstetrics, The American College of Obstetricians and Gynecologists. Practice bulletin no. 130: prediction and prevention of preterm birth. Obstet Gynecol. 2012 Oct;120(4):964-73. doi: 10.1097/AOG.0b013e3182723b1b. No abstract available. PMID 22996126
- [Background] Di Renzo GC, Giardina I, Clerici G, Mattei A, Alajmi AH, Gerli S. The role of progesterone in maternal and fetal medicine. Gynecol Endocrinol. 2012 Nov;28(11):925-32. doi: 10.3109/09513590.2012.730576. PMID 23057618
- [Background] Norwitz ER, Caughey AB. Progesterone supplementation and the prevention of preterm birth. Rev Obstet Gynecol. 2011 Summer;4(2):60-72. PMID 22102929
- [Background] Omar MH, Mashita MK, Lim PS, Jamil MA. Dydrogesterone in threatened abortion: pregnancy outcome. J Steroid Biochem Mol Biol. 2005 Dec;97(5):421-5. doi: 10.1016/j.jsbmb.2005.08.013. Epub 2005 Nov 15. PMID 16293412
- [Background] Carp H. A systematic review of dydrogesterone for the treatment of threatened miscarriage. Gynecol Endocrinol. 2012 Dec;28(12):983-90. doi: 10.3109/09513590.2012.702875. Epub 2012 Jul 16. PMID 22794306
- [Background] Queisser-Luft A. Dydrogesterone use during pregnancy: overview of birth defects reported since 1977. Early Hum Dev. 2009 Jun;85(6):375-7. doi: 10.1016/j.earlhumdev.2008.12.016. Epub 2009 Feb 3. PMID 19193503
- [Result] Dodd JM, Crowther CA, Cincotta R, Flenady V, Robinson JS. Progesterone supplementation for preventing preterm birth: a systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2005 Jun;84(6):526-33. doi: 10.1111/j.0001-6349.2005.00835.x. PMID 15901258
- [Result] Borna S, Sahabi N. Progesterone for maintenance tocolytic therapy after threatened preterm labour: a randomised controlled trial. Aust N Z J Obstet Gynaecol. 2008 Feb;48(1):58-63. doi: 10.1111/j.1479-828X.2007.00803.x. PMID 18275573
- [Result] Sharami SH, Zahiri Z, Shakiba M, Milani F. Maintenance therapy by vaginal progesterone after threatened idiopathic preterm labor: a randomized placebo-controlled double-blind trial. Int J Fertil Steril 2010;4:45-50.
- [Result] Arikan I, Barut A, Harma M, Harma IM. Effect of progesterone as a tocolytic and in maintenance therapy during preterm labor. Gynecol Obstet Invest. 2011;72(4):269-73. doi: 10.1159/000328719. Epub 2011 Nov 12. PMID 22086108
- [Result] Bomba-Opon DA, Kosinska-Kaczynska K, Kosinski P, Wegrzyn P, Kaczynski B, Wielgos M. Vaginal progesterone after tocolytic therapy in threatened preterm labor. J Matern Fetal Neonatal Med. 2012 Jul;25(7):1156-9. doi: 10.3109/14767058.2011.629014. Epub 2012 Apr 3. PMID 21967664
- [Result] Areia A, Fonseca E, Moura P. Progesterone use after successful treatment of threatened pre-term delivery. J Obstet Gynaecol. 2013 Oct;33(7):678-81. doi: 10.3109/01443615.2013.820266. PMID 24127952